CLINICAL TRIAL: NCT00942565
Title: Adjuvant Analgesic Effects of Low Dose Tramadol/Acetaminophen Combination After Open Gynaecological Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Chi Wai, Dr., The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 06-188 T/1213
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Postoperative Pain
Keywords: Open gynecological surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Ultracet; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Tramadol/acetaminophen (Active Comparator): The tramadol and acetaminophen combination was given to patients at the same day after surgery.
  Interventions: Drug: tramadol/acetaminophen
- acetaminophen (Active Comparator): Acetaminophen was used as active control.
  Interventions: Drug: acetaminophen

INTERVENTIONS:
Drug: tramadol/acetaminophen
  Arms: Tramadol/acetaminophen
Drug: acetaminophen
  Arms: acetaminophen

SUMMARY:
Patient experience moderate to severe pain after abdominal surgery. This post-operative pain can also contribute to complications such as respiratory impairment, cardiovascular events, ileus, sleep deprivation and mood disturbance. Opioid based patient-controlled analgesia (PCA) is commonly employed but opioids have the side effects such as respiratory depression, nausea and vomiting, sedation, pruritus and urinary retention. Bowel motility can also be affected. Consequently alternative or adjunct analgesic medications without these side-effects have been investigated in order to reduce opioid consumption.

Multimodal analgesia is a technique whereby a combination of analgesic drugs with different modes of action can be used to improve analgesia and decrease adverse effects by virtue of synergism. Postoperatively, with adjunctive analgesia, PCA morphine consumption as well as the side effects may be reduced. Non-steroidal anti-inflammatory drugs (NSAIDs) have been shown to be opioid sparing and decrease the adverse effects of PCA morphine. A recent review showed that acetaminophen combined with PCA could induce a significant opioid-sparing effect but the incidence of PCA morphine related side effects were not reduced.

It is common nowadays to give oral analgesic supplements to post-operative patients on PCA morphine. Tramadol, an analogue of codeine, is one of the choices. However, some of the patients cannot tolerate the side effects such as nausea, drowsiness, sweating, postural hypotension and dry mouth. Combination of tramadol 37.5 mg and acetaminophen 375 mg, which has been used successfully to treat post-operative pain, may improve analgesic response with better tolerability.

This study is to assess tramadol 37.5 mg and acetaminophen 375 mg combination on the efficacy of pain control, down stepping of morphine consumption and related adverse events with PCA use after open colorectal surgeries.

Objectives:

This study aims to compare and evaluate:

* The efficacy of tramadol/acetaminophen combination on postoperative pain relief after lower abdominal surgeries
* The effects of tramadol/acetaminophen combination on the consumption and the duration of PCA morphine use
* The adverse effects related to this regimen
* The effects on postoperative bowel function, tolerability of fluid and diet, ambulatory function, sleep, and duration of hospital stay
* The overall satisfaction of the patients

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled study.

Study site Patients will be recruited and studied at Queen Mary Hospital, Hong Kong.

Anaesthesia for operation No premedication will be prescribed. Patients will be induced with fentanyl 1 to1.5µg/kg, thiopentone 2-4mg/kg or propofol 2-3mg/kg and rocuronium 1mg/kg. Anaesthesia will be maintained with cisatracurium and isoflurane with air and oxygen. Intravenous morphine will be used for pain relief intraoperatively.

Postoperative PCA settings

After the operation, at the recovery area, patients will be given boluses of intravenous morphine until satisfactory pain control, i.e. numerical rating scale (NRS) less than 4. PCA machine will then be connected and patient will learn the technique of using PCA. The PCA pump will be programmed as follow:

Each bolus: 1 to 1.5mg Lockout interval: 5 minutes Maximum hourly dose limit: 0.1mg/kg for patients up to 65 years old and 0.075mg/kg for patients over 65 No background morphine infusion will be given. Intramuscular pethidine 0.5mg/kg four-hourly will be prescribed as rescue pain medications. Patients will be assessed everyday by the pain team of the hospital.

Randomisation and blinding

Patients will be randomised to one of the following 2 groups:

Group T: Tramadol 37.5mg / acetaminophen 325mg: 1 tablet 3 times daily orally Group P: Acetaminophen 500mg 3 times daily A computer-generated random sequence will decide the allocation order. The appearance of acetaminophen looks similar to the tramadol/acetaminophen combination. Both pain team members and patients will be blinded to the study medications. The study medications will be used for 48 hours after operation.

Follow-up and assessments Patients will be assessed each morning by the pain team. The daily average pain score at rest and during cough will be recorded in numerical rating scale (NRS). Average daily pain intensity (0=none, 1=mild, 2=moderate, 3=severe) and average daily relief (4=complete relief, 3=a lot, 2=moderate, 1=slight, 0=no, -1=worse pain) will be assessed. The tries/good ratio shown on PCA machine and the total amount of morphine used, daily rescue pain drug consumption will be charted. The adverse effects (nausea, vomiting, pruritus, dizziness, and others) will be recorded with their frequencies and severity graded. Sedation will be assessed based on the scale shown.

The ambulatory function, tolerability of fluid and diet and bowel function will also be assessed. Sleeping quality will be evaluated using NRS and reason for it asked.

The PCA machine will be off if the NRS pain score on cough is less than 4. Patients will then grade their overall satisfaction of pain relief at postoperative day 3.

Data Collection

Efficacy

* Resting and coughing NRS pain scores,
* Average daily pain intensity and average daily relief
* Tries/good ratio, cumulative morphine consumption,
* Rescue pain drug consumption every day until 2 days after stopping PCA
* Overall patient's satisfaction using NRS

Safety

- Adverse effects and their severity, sedation, ambulatory function, tolerability of fluid and diet, bowel function, and sleeping quality every day until off PCA

Demographics

* Age
* Sex
* Body weight
* ASA grading
* Operation duration
* Intraoperative opioids
* Morphine consumption at recovery room

ELIGIBILITY:
Inclusion Criteria:

* ASA I to III
* Age 18 to 80 years
* Scheduled for elective lower abdominal surgery (gynecological or colorectal surgery) at Queen Mary Hospital, Hong Kong

Exclusion Criteria:

* Allergy to tramadol, acetaminophen, or other opioid drugs
* Patient with epilepsy or history of seizures
* Concurrent use of selective serotonin uptake inhibitors, tricyclic antidepressants, or monoamine oxidase inhibitors
* Impaired or retarded mental state
* Impaired renal function, defined as preoperative serum creatinine level over 120µmol/L
* Impaired hepatic function, defined as preoperative serum albumin level less than 30g/L
* Intraoperative use of clonidine or dexmedetomidine
* Patient requiring postoperative mechanical ventilation
* Difficulties in using patient-controlled analgesia
* Pregnancy
* Current or previous drug abuser
* Alcoholism
* Patient refusal

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pain score | Postoperative 48 hours

SECONDARY OUTCOMES:
postoperative morphine consumption, side effect, recovery, sleeping quality, satisfaction | Postoperative 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, The University of Hong Kong, Hong Kong, Hong Kong